CLINICAL TRIAL: NCT04689217
Title: Intrathecal Nalbuphine is a Comparable Safer Alternative to Fentanyl for Intraoperative Pain Management During Uterine Exteriorization in Cesarean Section. A Randomized Controlled Trial.
Brief Title: Intrathecal Nalbuphine is a Comparable Safer Alternative to Fentanyl for Intraoperative Pain Management During Uterine Exteriorization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N- 26 / 2020
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Pain, Acute
Keywords: intrathecal nalbuphine; intrathecal fentanyl; exteriorization of the uterus; cesarean section
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group F (Experimental): will receive intrathecal injection of 0.5% hyperbaric bupivacaine plus 0.5 ml fentanyl (25 μg)
  Interventions: Drug: intrathecal drug injection
- Group N (Experimental): will receive intrathecal injection of 0.5% hyperbaric bupivacaine plus 0.8 mg nalbuphine hydrochloride
  Interventions: Drug: intrathecal drug injection
- Group C (Placebo Comparator): will receive intrathecal injection of 0.5% hyperbaric bupivacaine plus 0.5 ml normal saline
  Interventions: Drug: intrathecal drug injection

INTERVENTIONS:
Drug: intrathecal drug injection — All patients will be put in the sitting position and lean forward. After sterilization, Dural puncture will be performed at L4-L5 interspace or L3-L4 with a 25 gauge Quincke spinal needle.
  The patients will be divided equally into 3 groups according to the additive (fentanyl, nalbuphine or placebo), and all patients will receive the local anesthetic dose of 0.5% heavy bupivacaine according to weight and height
  Other Names: spinal opioid injection

SUMMARY:
In case of cesarean section (CS) delivery, spinal anesthesia is the best anesthetic choice. It is simple to perform with rapid onset of anesthesia and lower incidence of failed block. Spinal anesthesia avoids the risk of aspiration, the neonatal depressant effect that may occur with general anesthesia (GA), and provides postoperative analgesia, however, spinal anesthesia has a lesser control on the level of blockade, may give insufficient visceral pain block and may be associated with nausea and vomiting especially during peritoneal traction, closure and uterine manipulation, exteriorization and rotation. A previous study reported nausea and vomiting in up to 70.5% patients in the spinal group while the incidence of moderate to severe pain was more frequent in exteriorized uterus patients.

Increasing the dosage of intrathecal local anesthetic may contribute to a decrease in the occurrence of intraoperative visceral pain, but at the cost of the risk and adverse effects of greater blockade.A variety of adjuvants have been used to prevent these disadvantages. The commonly used adjuvants include opioids; α2 stimulants such as clonidine and dexmedetomidine; NMDA receptor antagonist such as ketamine; GABA receptor agonists such as midazolam.

The added intrathecal opioids as fentanyl and nalbuphine to local anesthetics give a sufficient intraoperative visceral analgesia when they were used in C.S., with less sympathetic block and hemodynamic effect, and reduces the need for intraoperative analgesics with prolongation of postoperative analgesia.

Nalbuphine, a mixed agonist-antagonist opioid, has a potential to attenuate the mu-opioid effects and to enhance the kappa-opioid effects. It was synthesized attempting to produce analgesia without the undesirable side effects of mu agonist. Also, its combination with mu agonist opioids was tried by many researchers to decrease the incidence and severity of the common mu agonist side effects (respiratory depression, undesirable sedation, pruritus, bradycardia, nausea, vomiting and urinary retention), plus it can antagonize spinal induced shivering. Meanwhile, the benefits of both kappa and mu analgesia can be obtained.

Few studies compared the effects of intrathecal nalbuphine (opioid agonist-antagonist) and fentanyl (opioid agonist) as adjuvants to bupivacaine in spinal blocked for CS with variable results. However, they didn't compare their ability to control the visceral pain aggravated by uterine exteriorization in cesarean section under spinal anesthesia. This study will try to answer the question is nalbuphine effective enough in such scenario to be used routinely as a safer alternative to fentanyl, which is the opioid in common practice added to bupivacaine?

Aim of the study:

To compare the ability of the used doses in the study of intrathecal nalbuphine and intrathecal fentanyl to control the visceral pain aggravated by uterine exteriorization in cesarean section under spinal anesthesia

Objectives:

* To evaluate the visual analog scale (VAS) for visceral abdominal and shoulder pain every 5 minutes and the maximum score will be recorded for 30 minutes from the time of baby delivery.
* To calculate the total fentanyl used for VAS ⩾ 4

ELIGIBILITY:
Inclusion Criteria:

* forty-two female patients
* ASA physical status I or II,
* age between 20 and 45 years,
* weight between 60 and 100 kg
* height between 160 and 180 cm

Exclusion Criteria:

* ASA III or IV,
* patient refusal,
* hypotensive patients,
* infection at the site of injection,
* coagulopathy
* weight <60 and > 100 kg,
* anticoagulant medications,
* pre-existing neurological disease.
* uncooperative patients,
* cardiac disorder
* respiratory disorder
* allergy to local anesthetics.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cesarean section patients
Enrollment: 135 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
intraoperative pain control | 30 minutes after baby delivery
  - The visual analog scale (VAS) for visceral abdominal pain in all groups after uterine exteriorization.VAS from 0 to 10 with 0 equal no pain and 10 equal the severist pain ever

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Bogra J, Arora N, Srivastava P. Synergistic effect of intrathecal fentanyl and bupivacaine in spinal anesthesia for cesarean section. BMC Anesthesiol. 2005 May 17;5(1):5. doi: 10.1186/1471-2253-5-5. PMID 15904498
- [Background] Gauchan S, Thapa C, Prasai A, Pyakurel K, Joshi I, Tulachan J. Effects of intrathecal fentanyl as an adjunct to hyperbaric bupivacaine in spinal anesthesia for elective caesarean section. Nepal Med Coll J. 2014 Sep;16(1):5-8. PMID 25799801
- [Background] Pedersen H, Santos AC, Steinberg ES, Schapiro HM, Harmon TW, Finster M. Incidence of visceral pain during cesarean section: the effect of varying doses of spinal bupivacaine. Anesth Analg. 1989 Jul;69(1):46-9. PMID 2742167
- [Background] Alahuhta S, Kangas-Saarela T, Hollmen AI, Edstrom HH. Visceral pain during caesarean section under spinal and epidural anaesthesia with bupivacaine. Acta Anaesthesiol Scand. 1990 Feb;34(2):95-8. doi: 10.1111/j.1399-6576.1990.tb03050.x. PMID 2407045